CLINICAL TRIAL: NCT06814366
Title: The Effect of Music and White Noise on Patients' Anxiety and Pain During Surgery for Impacted Mandibular Third Molar: A Single-Blind Randomized Controlled Trial
Brief Title: The Effect of Music and White Noise on Patients' Anxiety and Pain During Surgery for Impacted Mandibular Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Mine ALKAYA KARAGOZ, principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AU-FD-OMFS-MAK-001
Record Dates: First submitted 2025-01-30; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Anxiety State; Pain
Keywords: tooth extraction; anxiety; white noise
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group music and white noise (Experimental): Group music and white noise listened to a preselected playlist played against a pre-prepared standard white noise through headphones that prevent ambient noise during the procedure. The playlist consisted of popular songs of the time. The patient could choose the music they wanted to listen to from the playlist using a hand-held tablet.
  Interventions: Other: music and white noise intervention
- group music only (Experimental): Group music listened to the same preselected playlist without white noise through noise-isolating headphones during the procedure. The patient could choose the music they wanted to listen to from the playlist using a hand-held tablet.
  Interventions: Other: music intervention
- group control (No Intervention): Group control listened to the natural ambient noise during the procedure.

INTERVENTIONS:
Other: music and white noise intervention — The experimental groups were played a combination of music and white noise through headphones that blocked ambient noise during the surgical procedure. A playlist consisting of the popular songs of the era was prepared in advance. The patient could choose the music they wanted to listen to from the playlist using a hand-held tablet.
  Arms: group music and white noise
Other: music intervention — The experimental groups were played music a through headphones that blocked ambient noise during the surgical procedure. A playlist consisting of the popular songs of the era was prepared in advance. The patient could choose the music they wanted to listen to from the playlist using a hand-held tablet.
  Arms: group music only

SUMMARY:
The goal of this clinical trial is to evaluate the effect of music and whitenoise on the anxiety and pain level of patients who had impacted third molars surgery. The main questions it aims to answer are:

* Does music and white noise have an effect on the patient's intraoperative pain/pressure/discomfort?
* Does music and white noise have an effect on the patient's anxiety level?

The researchers compared the music and white noise, music-only and ambient noise groups to see if there was an effect on anxiety and pain levels.

STAI-S form was applied to all participants before surgery. They marked their anxiety levels on the VAS scale. After the procedure, STAI-S form was applied and they marked the anxiety levels on the VAS scale. The pressure/pain level which they felt during the procedure was evaluated by VAS scale.

DETAILED DESCRIPTION:
Our study was carried out on 66 patients, who applied to Ankara University Department of Oral and Maxillofacial Surgery, suffering from impacted mandibular third molars.

Group white noise and music listened to a preselected playlist played against a pre-prepared standard white noise through headphones that prevent ambient noise during the procedure. The playlist consisted of popular songs of the time. The patient could choose the music they wanted to listen to from the playlist using a hand-held tablet.

Group music only listened to the same preselected playlist without white noise through noise-isolating headphones during the procedure. The patient could choose the music they wanted to listen to from the playlist using a hand-held tablet.

Group control listened to the natural ambient noise during the procedure.

Surgical Procedure:

All patients were given a mouthwash with chlorhexidine gluconate before the surgery. Before the procedure, Nervus Alveolaris inferior block anesthesia and buccal infiltrative anesthesia were performed with 2.5% articain hydrochloride (Ultracain D-S forte ampoule, Sanofi Aventis) containing 1/100,000 epinephrine as a local anesthetic solution. In all three groups, a mucoperiosteal triangular flap was raised to reach the bone. After removing a sufficient amount of bone, the tooth was removed from the socket using a bein elevator. The original position of the flap was preserved, and the wounds were closed primarily using an atraumatic silk suture.

Data Collection The State-Trait Anxiety Inventory-State (STAI-S FORM) was administered to the patients before and after the procedure. Marking was made on the form containing a visual analog scale (VAS) for anxiety levels before the procedure. Post-procedure anxiety levels and pain/pressure feelings were marked on a separate form containing a VAS scale, and the desire to have the procedure performed again (1=never, 2=maybe/not sure, 3=willing) was questioned.

ELIGIBILITY:
Inclusion Criteria:

* Patients who applied to our clinic for impacted wisdom teeth extraction from the start date of the study
* Patients without any diagnosed psychological disorder
* Patients who gave their own voluntary consent to the study
* Patients who had no medical history that could affect third molar surgery,

Exclusion Criteria:

* Patients who do not agree to volunteer.
* Patients with any diagnosed psychological disorder
* Patients with mental and physical disorders that may hinder cooperation
* Pregnancy or lactating,
* Antidepressant or anxiolytic drug use, having a disease that could prevent the surgery,
* A severe infection around the impacted third molar
* A prior tooth extraction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
STAI-S | preoperative and through the surgery is over, about an hour after the patient entered the operating room
  State anxiety measured on STAI-S (Spielberger State Anxiety Inventory). The total score can range from 20 to 80, with higher scores indicating more anxiety.
ANXIETY VAS | preoperative and through the surgery is over, about an hour after the patient entered the operating room
  Anxiety measured on a VAS (Visual Analog Scale). A closed-ended scale of 0-10 cm ("0" no anxiety, "10" maximum imaginable anxiety) was used in the study
PAIN VAS | perioperative
  Pain measured on a VAS (Visual Analog Scale ). A closed-ended scale of 0-10 cm ("0" no anxiety, "10" maximum imaginable anxiety) was used in the study

OTHER OUTCOMES:
willingness | through the surgery is over, about an hour after the patient entered the operating room
  The desire to undergo the surgical procedure again (1=never, 2=maybe/not sure, 3=willing) under the same conditions was questioned.

CONTACTS AND LOCATIONS:
Overall Officials: mine alkaya karagoz, DDS, Principal Investigator — Alanya Alaaddin Keykubat University
Locations (1):
- Ankara University, Ankara, Yenimahalle/ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YK, Kim SM, Myoung H. Musical intervention reduces patients' anxiety in surgical extraction of an impacted mandibular third molar. J Oral Maxillofac Surg. 2011 Apr;69(4):1036-45. doi: 10.1016/j.joms.2010.02.045. Epub 2010 Aug 12. PMID 20708320
- [Background] Song M, Li N, Zhang X, Shang Y, Yan L, Chu J, Sun R, Xu Y. Music for reducing the anxiety and pain of patients undergoing a biopsy: A meta-analysis. J Adv Nurs. 2018 May;74(5):1016-1029. doi: 10.1111/jan.13509. Epub 2017 Dec 21. PMID 29171070
- [Background] Ilkkaya NK, Ustun FE, Sener EB, Kaya C, Ustun YB, Koksal E, Kocamanoglu IS, Ozkan F. The effects of music, white noise, and ambient noise on sedation and anxiety in patients under spinal anesthesia during surgery. J Perianesth Nurs. 2014 Oct;29(5):418-26. doi: 10.1016/j.jopan.2014.05.008. PMID 25261145